CLINICAL TRIAL: NCT02984527
Title: Comparison of Skin Swaps From Traditional Bed Baths Versus Disposable Wet Wipes
Brief Title: Traditional Bed Baths Versus Disposable Wet Wipes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Hospital of Southern Jutland (Other)
Responsible Party: Principal Investigator, Pia Lysdal Veje, PhD student, University of Southern Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SDUSF-2015-65/R1 - (205)
Record Dates: First submitted 2016-11-29; First posted 2016-12-07 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Intimate Hygiene
MeSH Terms: interventions — Hydrotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- water and soap first day (Active Comparator): Intimate hygiene performed with water and soap first day and disposable wet wipes second day
  Interventions: Device: wet wipes; Device: water and soap
- disposable wet wipes first day (Active Comparator): Intimate hygiene performed with wet wipes first day and water and soap second day
  Interventions: Device: wet wipes; Device: water and soap

INTERVENTIONS:
Device: wet wipes — intimate hygiene with disposable wet wipes
Device: water and soap — Intimate hygiene with water and soap

SUMMARY:
The Purpose of the study is to compare the effectiveness on microbiological counts from skin swaps after wash with water and soap or wet wipes.

DETAILED DESCRIPTION:
The study is a crossover clinical trial where the effect of two interventions is compared on the same subject.

The two interventions are:

* Intimate hygiene with water and soap
* Intimate hygiene with prepackaged disposable wet wipes

Null hypothesis: Same effectiveness to reduce microbiological counts on skin

Alternative hypothesis: Significant different effectiveness to reduce microbiological counts on skin

Each individual receives the two interventions in random order. The effect of the interventions on microbiological counts on the patients skin is evaluated on the same patient.

A crossover trial requires half the number of participants and reduces confounding factors.

All participants receive a sequence of the two different interventions. But there is a sufficient gab between the two interventions to ensure a washout period and avoid a crossover effect. In this study this is 12-24 hours.

The study uses block randomization, without intra block correlation to achieve allocation balance over time.

Furthermore it may prevent some predictable allocation.

Microbiological sampling with moistened swaps and aseptic techniques, sterile equipment and sterile recovery medium (Stewarts Medium) are used to obtain skin samples from the patients before and after intimate hygiene with water and soap and wet wipes.

Differences in microbiological skin counts will be compared (delta values) before and after the two interventions and between interventions.

Data will be blinded during microbiological count and statistical analyses.

Analyses:

Data are structured in CASTOR and will be stored in a secure Team Collaboration Software Tool (SharePoint).

Descriptive analysis including mean, median, confidence interval, standard deviation, and standard error.

Statistical analyses will be performed using STATA. Test of differences will be performed by simple t- test or Wilcoxon sign rank test, depending on the distribution of the data. A multiple regression analysis including possible confounders will be considered.

Inclusion of 68 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients who need intimate hygiene
* Admitted for minimum two days
* Understand oral information
* And apple to sign written consent

Exclusion Criteria:

* Diarrhea
* Dementia
* Dying

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
microbiological counts on skin before and after interventions | two consecutive days
  microbiological counts from skin swaps before and after washing with water and soap and before and after washing with disposable wipes

CONTACTS AND LOCATIONS:
Overall Officials: Jette Primdahl, PhD, Study Chair — Hospital of Southern Jutland
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No